CLINICAL TRIAL: NCT02901275
Title: Using Dronabinol to Enhance the Analgesic Effect of Hydromorphone in Humans
Brief Title: Enhancing Medication-based Analgesia in Humans
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: Triple | Purpose: Basic Science
Other Study IDs: IRB00097937
Record Dates: First submitted 2016-07-28; First posted 2016-09-15 (Estimated); Results first posted 2021-06-07 (Actual); Last update posted 2023-11-07 (Actual); Status verified 2023-11

CONDITIONS: Pain; Cannabis; Opioid Use, Unspecified
Keywords: Clinical Trial, Phase II; Analgesia; Abuse Potential
MeSH Terms: conditions — Pain; Marijuana Abuse; Agnosia

STUDY DESIGN:
Intervention Model Description: Each participant completed each of the 5 study conditions (identified here as arms).
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- Placebo + Placebo (Placebo Comparator): Within-subject double-blind, double-dummy administration of placebo + placebo. Order of dose randomized session days 2-5.
  Interventions: Drug: Within-subject test of blinded study medications
- Hydromorphone (oral) 4mg + Placebo (Active Comparator): Within-subject double-blind, double-dummy administration of hydromorphone (oral) 4mg + placebo. Always administered during session 1.
  Interventions: Drug: Within-subject test of blinded study medications
- Hydromorphone (oral) 4mg / Dronabinol (oral) 2.5mg (Experimental): Within-subject double-blind, double-dummy administration of hydromorphone (oral) 4mg + dronabinol (oral) 2.5mg. Order of dose randomized session days 2-5.
  Interventions: Drug: Within-subject test of blinded study medications
- Hydromorphone (oral) 4mg / Dronabinol (oral) 5mg (Experimental): Within-subject double-blind, double-dummy administration of hydromorphone (oral) 4mg + dronabinol (oral) 5.0mg. Order of dose randomized session days 2-5.
  Interventions: Drug: Within-subject test of blinded study medications
- Hydromorphone (oral) 4mg / Dronabinol (oral) 10mg (Experimental): Within-subject double-blind, double-dummy administration of hydromorphone (oral) 4mg + dronabinol (oral) 10mg. Order of dose randomized session days 2-5 but was never the first hydromorphone 4mg + dronabinol combination dose.
  Interventions: Drug: Within-subject test of blinded study medications

INTERVENTIONS:
Drug: Within-subject test of blinded study medications — Within-subject double-blind, double-dummy, study design wherein all participants received all doses in 8-hour outpatient sessions. Primary outcomes assessed during 8-hour outpatient sessions and included laboratory pain testing, subjective reports of drug effects, and cognitive performance, evaluated as a function of study medication condition.

SUMMARY:
This is a single-group, within-subject, double-blind, double-dummy, placebo and active-controlled study evaluated whether the FDA-approved cannabinoid dronabinol (Marinol) would enhance analgesia, subjective reports, and cognitive performance when compared to the FDA-approved opioid hydromorphone (Dilaudid).

DETAILED DESCRIPTION:
This was a human laboratory systematic examination of whether adding the FDA-approved cannabinoid dronabinol (Marinol; oral) to the FDA-approved opioid hydromorphone (Dilaudid; oral) would change the experience of hydromorphone as rated by laboratory measures of pain, subjective reports of drug effects, and cognitive performance. Subjects are healthy individuals with no history of drug use disorder. Study subjects and staff were completed blinded to the study drugs and the class of drugs under investigation and were informed that subjects may receive opioids, stimulants, cannabinoids, benzodiazepines, over the counter medications, and/or placebo. All participants completed all sessions. Sessions lasted up to 8-hours and were conducted at least 7 days apart on an outpatient basis. Primary outcomes were collected from participants prior to dosing and at several hour periods post-dosing.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18-75
* Urine sample tests negative for common illicit substances of abuse, including cannabis
* Medically cleared to take study medications
* Are not pregnant or breast feeding
* Willing to comply with the study protocol.

Exclusion Criteria:

* Meet DSM-5 criteria for alcohol/substance use disorder
* Taking opioids for pain
* Previous adverse reaction to a cannabinoid product
* Prescribed and taking stimulants or benzodiazepines
* Answer "yes" to item 1 of the Brief Pain Inventory indicating chronic pain
* Self-report any illicit drug use in the past 7 days
* Presence of any clinically significant medical/psychiatric illness judged by the investigators to put subject at elevated risk for experiencing an adverse event
* History of seizure disorder
* Have a known allergy to the study medications or sesame seed oil
* Taking medications contraindicated with hydromorphone or dronabinol
* Have a history of clinically significant cardiac arrhythmias or vasopastic disease
* Have an abnormal and clinically-significant ECG

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2016-12 (Actual); Primary Completion 2020-03-23 (Actual); Study Completion 2020-03-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kelly Dunn, PhD, Principal Investigator — Principal Investigator; Claudia Campbell, PhD, Principal Investigator — Principal Investigator
Locations (1):
- Johns Hopkins University, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This is a within-subject study, and all participants (n=29) completed all study conditions. The same 29 participants moved from one treatment arm to the next.
Groups:
- Full Participant Sample: Each participant completed the following five study conditions (arms) in randomized order:
  Placebo + Placebo condition
  Hydromorphone (oral) 4mg + placebo condition
  Hydromorphone (oral) 4mg + Dronabinol (oral) 2.5mg condition
  Hydromorphone (oral) 4mg + Dronabinol (oral) 5mg condition
  Hydromorphone (oral) 4mg + Dronabinol (oral) 10mg condition
Period: Overall Study
Arm/Group | Full Participant Sample
Started | 29
Placebo + Placebo | 29
Hydromorphone (Oral) 4mg + Placebo | 29
Hydromorphone (Oral) 4mg + Dronabinol (Oral) 2.5mg | 29
Hydromorphone (Oral) 4mg + Dronabinol (Oral) 5mg | 29
Hydromorphone (Oral) 4mg + Dronabinol (Oral) 10mg | 29
Completed | 29
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- All Participants: This is a within group study and same participants went through all treatment arms.
Arm/Group | All Participants
Number analyzed (Participants) | 29
Age, Continuous [Mean (Standard Deviation); unit: years] | 30.4 (9.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15
  Male | 14
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 27
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 3
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 12
  White | 14
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 29

OUTCOME MEASURES:

1. Primary Outcome: Mean Change From Baseline in Seconds to Withdraw Hand From Cold Pressor Laboratory Pain Task
Description: Compare study conditions in seconds to withdraw hand from cold pressor laboratory pain task, where longer time periods reflect higher tolerance to pain.
Time Frame: Baseline and time of hand withdrawal from cold pressor, up to 60 seconds
Measure: Mean (Standard Error); unit: seconds
Groups:
- Placebo + Placebo Condition: Within-subject placebo + placebo control condition.
- Hydromorphone (Oral) 4mg + Placebo Condition: Within-subject hydromorphone 4mg + placebo control condition.
- Hydromorphone (Oral) 4mg + Dronabinol (Oral) 2.5mg: Within-subject hydromorphone 4mg+ dronabinol 2.5mg experimental condition
- Hydromorphone (Oral) 4mg + Dronabinol (Oral) 5.0mg: Within-subject hydromorphone 4mg+ dronabinol 5.0mg experimental condition
- Hydromorphone (Oral) 4mg + Dronabinol (Oral) 10mg: Within-subject hydromorphone 4mg+ dronabinol 10mg experimental condition
Arm/Group | Placebo + Placebo Condition | Hydromorphone (Oral) 4mg + Placebo Condition | Hydromorphone (Oral) 4mg + Dronabinol (Oral) 2.5mg | Hydromorphone (Oral) 4mg + Dronabinol (Oral) 5.0mg | Hydromorphone (Oral) 4mg + Dronabinol (Oral) 10mg
Number analyzed (Participants) | 29 | 29 | 29 | 29 | 29
seconds | 25.4 (12.7) | 33.9 (15.7) | 31.7 (10.9) | 36.7 (12.6) | 18.1 (5.4)
Statistical Analysis 1: Comparison: Placebo + Placebo Condition vs Hydromorphone (Oral) 4mg + Placebo Condition vs Hydromorphone (Oral) 4mg + Dronabinol (Oral) 2.5mg vs Hydromorphone (Oral) 4mg + Dronabinol (Oral) 5.0mg vs Hydromorphone (Oral) 4mg + Dronabinol (Oral) 10mg; Test type: Superiority; p = 0.61, Mixed Models Analysis — No covariate or correction for multiple comparisons. a priori statistical threshold is p<.05

2. Primary Outcome: Mean Peak Rating of "Drug Effect" (0-100) as Measured by the Visual Analog Rating Scale
Description: Mean peak of Visual Analog Scale ratings of Drug Effect (0-100) compared across each study condition, with higher ratings reflecting stronger drug effects.
Time Frame: 8-hour study session
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo + Placebo Condition | Hydromorphone (Oral) 4mg + Placebo Condition | Hydromorphone (Oral) 4mg + Dronabinol (Oral) 2.5mg | Hydromorphone (Oral) 4mg + Dronabinol (Oral) 5.0mg | Hydromorphone (Oral) 4mg + Dronabinol (Oral) 10mg
Number analyzed (Participants) | 29 | 29 | 29 | 29 | 29
score on a scale | 10.0 (10.1) | 51.1 (22.9) | 55.7 (29.4) | 55.7 (29.3) | 56.9 (31.7)
Statistical Analysis 1: Comparison: Placebo + Placebo Condition vs Hydromorphone (Oral) 4mg + Placebo Condition vs Hydromorphone (Oral) 4mg + Dronabinol (Oral) 2.5mg vs Hydromorphone (Oral) 4mg + Dronabinol (Oral) 5.0mg vs Hydromorphone (Oral) 4mg + Dronabinol (Oral) 10mg; Test type: Superiority; p < .0001, Mixed Models Analysis — No covariates or correction for multiple comparisons. a priori threshold is p<.05

3. Primary Outcome: Mean Change From Baseline in Maximum Percent Correct on Digit Symbol Substitution Test of Cognitive Behavior
Description: Within-subject comparison of study conditions on the Digit Symbol Substitution Test (DSST), a measure of cognitive performance that is sensitive to drug effects, wherein lower percent scores reflect worse performance and suggest greater drug-related impairment.
Time Frame: Baseline and 8-hours
Measure: Mean (Full Range); unit: Mean Percent Correct
Arm/Group | Placebo + Placebo Condition | Hydromorphone (Oral) 4mg + Placebo Condition | Hydromorphone (Oral) 4mg + Dronabinol (Oral) 2.5mg | Hydromorphone (Oral) 4mg + Dronabinol (Oral) 5.0mg | Hydromorphone (Oral) 4mg + Dronabinol (Oral) 10mg
Number analyzed (Participants) | 29 | 29 | 29 | 29 | 29
Mean Percent Correct | 10.2 [0 to 100] | 5.1 [0 to 100] | 10.1 [0 to 100] | 10.3 [0 to 100] | 3.6 [0 to 100]
Statistical Analysis 1: Comparison: Placebo + Placebo Condition vs Hydromorphone (Oral) 4mg + Placebo Condition vs Hydromorphone (Oral) 4mg + Dronabinol (Oral) 2.5mg vs Hydromorphone (Oral) 4mg + Dronabinol (Oral) 5.0mg vs Hydromorphone (Oral) 4mg + Dronabinol (Oral) 10mg; Test type: Superiority; p = 0.51, Mixed Models Analysis — No covariate or correction for multiple comparisons. a priori threshold for significance is p<.05

ADVERSE EVENTS:
Time Frame: Adverse events were documented throughout each of the 5 outpatient, 8-hour sessions, up to 40 hours.
Description: Adverse events were prompted systematically each hour throughout the session and documented according to good clinical practices. Spontaneously reported adverse events were also documented. All reports of symptoms were categorized as discrete events, such that one experience that included more than 1 symptom would be represented by more than 1 event. Events reported here were all rated as definitely or possibly related to study medication, collapsed across severity (mild, moderate, or severe).
Arm/Group | Placebo + Placebo Condition | Hydromorphone (Oral) 4mg + Placebo Condition | Hydromorphone (Oral) 4mg + Dronabinol (Oral) 2.5mg | Hydromorphone (Oral) 4mg + Dronabinol (Oral) 5.0mg | Hydromorphone (Oral) 4mg + Dronabinol (Oral) 10mg
All-Cause Mortality (participants affected / at risk) | 0/29 | 0/29 | 0/29 | 0/29 | 0/29
Serious Adverse Events (participants affected / at risk) | 0/29 | 0/29 | 0/29 | 0/29 | 0/29
Other Adverse Events (participants affected / at risk) | 12/29 | 22/29 | 11/29 | 25/29 | 21/29
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo + Placebo Condition (N=29) | Hydromorphone (Oral) 4mg + Placebo Condition (N=29) | Hydromorphone (Oral) 4mg + Dronabinol (Oral) 2.5mg (N=29) | Hydromorphone (Oral) 4mg + Dronabinol (Oral) 5.0mg (N=29) | Hydromorphone (Oral) 4mg + Dronabinol (Oral) 10mg (N=29)
Headache (Blood and lymphatic system disorders) | 2 (2) | 2 (2) | 3 (3) | 0 (0) | 0 (0)
Malaise (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Angina (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
Appetite- Increased (Gastrointestinal disorders) | 3 (3) | 3 (3) | 2 (2) | 6 (6) | 3 (3)
Dry Mouth (Gastrointestinal disorders) | 2 (2) | 2 (2) | 3 (3) | 9 (9) | 9 (9)
Epigastric Discomfort (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Nausea (Gastrointestinal disorders) | 2 (2) | 8 (8) | 7 (7) | 8 (8) | 11 (11)
Vomiting (Gastrointestinal disorders) | 0 (0) | 7 (7) | 1 (1) | 8 (8) | 2 (2)
Light Headedness (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Agitation (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Delerium (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Depression (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Dizziness (Nervous system disorders) | 2 (2) | 3 (3) | 3 (3) | 5 (5) | 2 (2)
Fatigue (Nervous system disorders) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Hypersomnia (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Impaired- Groggy (Nervous system disorders) | 5 (5) | 3 (3) | 3 (3) | 8 (8) | 8 (8)
Lethargy (Nervous system disorders) | 0 (0) | 3 (3) | 2 (2) | 2 (2) | 2 (2)
Light Headed (Nervous system disorders) | 0 (0) | 1 (1) | 3 (3) | 0 (0) | 0 (0)
Nervousness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Paranoid (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Parasthesia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Restlessness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Shaky (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Hyperventilation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rhinitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Photosensitivity (Eye disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Blurred Vision (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 1 (1)
Hot Flashes (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 2 (2)
Lacrimation (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Panic Attack (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Drowsiness (Nervous system disorders) | 12 (12) | 22 (22) | 11 (11) | 25 (25) | 21 (21)
Euphoria (Nervous system disorders) | 0 (0) | 9 (9) | 11 (11) | 18 (18) | 13 (13)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-02-12): https://cdn.clinicaltrials.gov/large-docs/75/NCT02901275/Prot_SAP_002.pdf
  • Informed Consent Form (2017-11-13): https://cdn.clinicaltrials.gov/large-docs/75/NCT02901275/ICF_001.pdf